CLINICAL TRIAL: NCT03348085
Title: Taipei Tzu Chi Hospital , Buddhist Tzu Chi Medical Foundation
Brief Title: Is Optimal Minute Ventilation a Predictor of Weaning in Patients With Prolong Mechanical Ventilation?
Status: Completed | Type: Observational
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 04-XD25-067
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2016-01

CONDITIONS: Chronic Respiratory Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention.

SUMMARY:
1. purpose of study: optimal minute could be the prediction of successful weaning and become the new weaning parameter.
2. study design: inclusion criteria: investigators will perform this study at our respiratory care center. Patients who had been maintained on mechanical ventilator in excess of 3 weeks before respiratory care center admission and all previous weaning attempts had ailed.

   Exclusion criteria: Patients do not have spontaneous breath. Terminal cancer stage and unstable hemodynamics condition.
3. study duration: 2016/01/01~12/31

DETAILED DESCRIPTION:
Investigators will preform this study at our respiratory care center. Initially, Investigators collected all physiological parameters and baseline characteristics of patients with prolong mechanical ventilator. Investigators use Gold-Galileo ventilator and patients use adaptive support ventilation mode. In adaptive support ventilation, the clinician enters a target minute volume , using a parameter called minute ventilation percentage. The minute ventilation percentage setting be initially set at 100% (the 100%minute ventilation setting), which provides a target minute ventilation of 0.1 L/min/kg of ideal body weight . Investigators observed respiratory frequency of patients, the minute ventilation percentage was increased every 5 min until the mandatory breath began to appear and spontaneous rate is zero. If the minute ventilation percentage had exceeded 250%, but patients do not have mandatory rate appeared, the optimal minute ventilation of the patient is means above 250%. Investigators also measure other weaning parameters. Finally, Investigators analyze the prediction of optimal minute ventilation as a weaning parameter.

ELIGIBILITY:
Inclusion Criteria:

* patients who had been maintained on mechanical ventilation in excess of 3 weeks before respiratory care center admission and all previous weaning attempts had failed.

Exclusion Criteria:

* Patients do not have spontaneous breath. Patients do not use invasive mechanical ventilator. Terminal cancer stage and hemodynamics unstable.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients are included in this study if they had been maintained on mechanical ventilation in excess of 3 weeks before respiratory care center admission, and all previous weaning attempts had failed.
  Patients are eligible for respiratory care center admission : hemodynamics stability, no vasoactive drug infusion for 24 hours or more before transfer, stable oxygen requirements(FIO2<40%,PERP<10 cmH2O), no hepatic failure, no requirement for surgical intervention within the 2 weeks, .
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
The prediction of optimal minute ventilation as successful weaning parameters in patients with prolong mechanical ventilator. | 2016/01/01~2016/12/31,1 year
  Investigators observed the condition of patients with adaptive spontaneous ventilation mode that the patient admitted to respiratory care center first day

CONTACTS AND LOCATIONS:
Overall Officials: YaRu Liang, Study Chair — Taipei Tzuchi hospital , Buddhist Tzu chi medical foundation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ntoumenopoulos G. Rehabilitation during mechanical ventilation: Review of the recent literature. Intensive Crit Care Nurs. 2015 Jun;31(3):125-32. doi: 10.1016/j.iccn.2015.02.001. Epub 2015 May 27. PMID 26026495
- [Background] MacIntyre NR, Epstein SK, Carson S, Scheinhorn D, Christopher K, Muldoon S; National Association for Medical Direction of Respiratory Care. Management of patients requiring prolonged mechanical ventilation: report of a NAMDRC consensus conference. Chest. 2005 Dec;128(6):3937-54. doi: 10.1378/chest.128.6.3937. PMID 16354866
- [Background] King C, Moores LK. Controversies in mechanical ventilation: when should a tracheotomy be placed? Clin Chest Med. 2008 Jun;29(2):253-63, vi. doi: 10.1016/j.ccm.2008.01.002. PMID 18440435
- [Background] Scheinhorn DJ, Artinian BM, Catlin JL. Weaning from prolonged mechanical ventilation. The experience at a regional weaning center. Chest. 1994 Feb;105(2):534-9. doi: 10.1378/chest.105.2.534. PMID 8306758
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Frutos-Vivar F, Esteban A. Critical illness polyneuropathy: a new (or old?) reason for weaning failure. Crit Care Med. 2005 Feb;33(2):452-3. doi: 10.1097/01.ccm.0000153525.37281.d4. No abstract available. PMID 15699857
- [Background] Wu YK, Tsai YH, Lan CC, Huang CY, Lee CH, Kao KC, Fu JY. Prolonged mechanical ventilation in a respiratory-care setting: a comparison of outcome between tracheostomized and translaryngeal intubated patients. Crit Care. 2010;14(2):R26. doi: 10.1186/cc8890. Epub 2010 Mar 1. PMID 20193057
- [Background] Schonhofer B. [Effect on the duration of mechanical ventilation of identifying patients capable of breathing spontaneously]. Pneumologie. 1997 Jun;51(6):599-600. No abstract available. German. PMID 9333795
- [Background] Verceles AC, Diaz-Abad M, Geiger-Brown J, Scharf SM. Testing the prognostic value of the rapid shallow breathing index in predicting successful weaning in patients requiring prolonged mechanical ventilation. Heart Lung. 2012 Nov-Dec;41(6):546-52. doi: 10.1016/j.hrtlng.2012.06.003. Epub 2012 Jul 6. PMID 22770598
- [Background] Wu CP, Lin HI, Perng WC, Yang SH, Chen CW, Huang YC, Huang KL. Correlation between the %MinVol setting and work of breathing during adaptive support ventilation in patients with respiratory failure. Respir Care. 2010 Mar;55(3):334-41. PMID 20196884
- [Background] OTIS AB, MCKERROW CB, BARTLETT RA, MEAD J, MCILROY MB, SELVER-STONE NJ, RADFORD EP Jr. Mechanical factors in distribution of pulmonary ventilation. J Appl Physiol. 1956 Jan;8(4):427-43. doi: 10.1152/jappl.1956.8.4.427. No abstract available. PMID 13286206